CLINICAL TRIAL: NCT05963165
Title: Early Speech Therapy Using Non-phonatory Exercises in Patients with Unilateral Vocal Fols Paralysis After Thyroidectomy: a Randomized Clinical Trial
Brief Title: Non-phonatory Exercises in Patients with Unilateral Vocal Fold Paralysis Post-thyroidectomy
Acronym: ENFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D'Alatri Lucia, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5559
Record Dates: First submitted 2023-07-04; First posted 2023-07-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2023-07

CONDITIONS: Unilateral Vocal Cord Paralysis
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients who will perform non-phonatory exercises in parallel with medical therapy for the first week
  Interventions: Behavioral: Non-phonatory exercises
- Control group (No Intervention): patients who will perform standard medical therapy only during the first week.

INTERVENTIONS:
Behavioral: Non-phonatory exercises — Muscle exercises that favor glottic adduction without vocal emissions
  Arms: Experimental group

SUMMARY:
Thyroidectomy is the most common iatrogenic cause of vocal fold paralysis. Patients complain of hoarseness caused by incomplete glottic closure and have effort to raise vocal intensity with consequent elevation of the larynx and/or involvement of supraglottic structures in phonation. These compensation mechanisms result in a shift of the fundamental frequency towards more serious tones or falsetto voice emissions.

The first choice treatment is speech therapy which aims to obtain better glottic closure, preventing ankylosis of the crico-arytenoid joint. In order to promote better glottic closure without risking the onset or increase of dysfunctional compensation, the idea behind this project is to propose non-phonatory adduction exercises in the first post-operative week.

The primary objective of the study is to compare patients who will perform non-phonatory exercises in parallel with medical therapy for one week and patients who will perform standard medical therapy only during the first week.

ELIGIBILITY:
Inclusion Criteria:

* vocal fold paralysis after thyrodectomy
* ability to sign an informed consent

Exclusion Criteria:

* Vocal fold paralysis with different etiology
* Previous history of laryngeal, pulmonary or gastric surgery
* History of vocal or laryngeal pathologies that have required therapy
* Current or previous lung disorders
* Hearing loss
* Motor or neurological deficits
* Presence of malignant diseases
* Presence of speech or reading disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Degree of glottic closure | 3 months
  A videostrobolaryngoscopy will be performed. The recorded videos will be viewed by expert clinicians and a numerical score will be assigned relating to the degree of glottic adduction on a 7-point scale.

SECONDARY OUTCOMES:
Acoustic analysis (fundamental frequency) | 3 months
  Through the use of the "Praat" software, on the reading of the piece "The desert" and on a sustained /a/ the Fundamental Frequency (F0, Hz) will be analysed.
Acoustic analysis (NHR) | 3 months
  Through the use of the "Praat" software, on the reading of the piece "The desert" and on a sustained /a/ the noise/harmonics ratio (NHR) will be analysed.
Acoustic analysis (Jitter%) | 3 months
  Through the use of the "Praat" software, on the reading of the piece "The desert" and on a sustained /a/ the Jitter (%) will be analysed.
Acoustic analysis (Shimmer%) | 3 months
  Through the use of the "Praat" software, on the reading of the piece "The desert" and on a sustained /a/ the Shimmer ( %) will be analysed.
  f
Acoustic analysis (Flow) | 3 months
  Through the use of the "Praat" software, on the reading of the piece "The desert" and on a sustained /a/ the minimum frequency (Flow) will be analysed.
Acoustic analysis (Fhigh) | 3 months
  Through the use of the "Praat" software, on the reading of the piece "The desert" and on a sustained /a/ the maximum frequency (Fhigh) will be analysed.
Acoustic analysis (intensity) | 3 months
  Through the use of the "Praat" software, on the reading of the piece "The desert" and on a sustained /a/ the intensity (dB) will be analysed.
MPT | 3 months
  the Maximum Phonatory Time (MPT) will be evaluated on a sustained /a/ (minimum 3 seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - IRCCS, Roma, Italy, Italy